CLINICAL TRIAL: NCT02496143
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral Administration of EC-18 in Healthy Subjects
Brief Title: A Safety and PK Study of EC-18 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EC-18-001
Record Dates: First submitted 2015-06-29; First posted 2015-07-14 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Healthy Volunteers; Phase I; Placebo controlled; Single Ascending Dose; PK; Oral administration; Softgel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 500 mg EC-18 dose or placebo
  Interventions: Drug: EC-18; Drug: Placebo
- Cohort 2 (Experimental): 1000 mg EC-18 dose orplacebo
  Interventions: Drug: EC-18; Drug: Placebo
- Cohort 3 (Experimental): 2000 mg EC-18 dose or placebo
  Interventions: Drug: EC-18; Drug: Placebo
- Cohort 4 (Experimental): 4000 mg EC-18 dose or placebo
  Interventions: Drug: EC-18; Drug: Placebo

INTERVENTIONS:
Drug: EC-18 — EC-18 will be supplied as 500 mg Softgel capsules. The study will include up to four sequential dose cohorts. Six subjects in each cohort will be randomized to receive EC-18: 500, 1000, 2000, or 4000 mg by oral administration of 1, 2, 4, and 8 EC-18 capsules, for Cohorts 1, 2, 3 or 4, respectively.
  Other Names: EC-18 Softgel capsule
Drug: Placebo — Placebo will be supplied as Softgel capsules. The study will include up to four sequential dose cohorts. Two subjects in each cohort will be randomized to placebo and will receive 1, 2, 4 or 8 placebo capsules for Cohorts 1, 2, 3 or 4, respectively.

SUMMARY:
The purpose of this study is to determine if EC-18 is safe and tolerable in healthy subjects.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled study of the safety, tolerability, PK, and pharmacodynamics of single ascending doses of EC-18 or placebo. If no dose limiting toxicity (DLT) is observed in Cohort One, the dose of EC-18 will be increased to in Cohorts Two, Three, and Four, respectively. Dose escalation to each successive cohort of subjects will not occur until a review of the safety and tolerability data from the previous cohort is completed and the Investigator, Sponsor, and study Medical Monitor together confirm the safety and tolerability of EC-18 given at that dose level.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential must use an acceptable birth control method throughout the study and for 14 days after the dose of study drug.
* Females of non-childbearing potential (defined as surgically sterilized [tubal ligation/hysterectomy/bilateral salpingo-oophorectomy] or postmenopausal for >2 years) with a negative urine human chorionic gonadotropin pregnancy test at the Screening Visit.
* Males willing to practice contraception (condom + spermicide) during the study and for 14 days after completion of the study, or who have a female partner using barrier or oral contraception during that timeframe.
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive.
* Ability to understand and give informed consent and provide authorization for use of protected health information (Health Insurance Portability and Accountability Act).
* Willing and able to be confined to the research clinic as required by the protocol.

Exclusion Criteria:

* Febrile (temperature ≥99.5°F/37.5°C) at the Screening Visit or at admission to the research clinic on Day -1.
* Clinically significant laboratory findings at the Screening Visit defined as the following:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin >1.5 x upper limit of normal (ULN)
  * Blood urea nitrogen (BUN), creatinine >1.25 x ULN
  * White blood cell (WBC) count <0.9 x lower limit of normal (LLN) or >1.1 x ULN
  * Hemoglobin or hematocrit <0.9 x LLN or >1.1 x ULN
  * Platelet count <0.9 x LLN or >1.1 x ULN
  * Glucose <0.9 x LLN or >1.25 x ULN
  * Thyroid-stimulating hormone (TSH) <0.75 x LLN or >1.25 x ULN or any other laboratory, ECG, vital sign, or physical abnormality that, in the investigator's opinion, unfavorably increases the risk of study participation.
* Positivity for human immunodeficiency virus (HIV) or receiving active antiretroviral therapy, hepatitis B surface antigen positivity, or hepatitis C positivity.
* History of drug or alcohol abuse within the past 2 years.
* Females who are pregnant or intend to get pregnant over the next month.
* Positive urine pregnancy test at the Screening Visit or at admission to the research clinic on Day -1.
* Positive urine drug or breath alcohol test at the Screening Visit or at admission to the research clinic on Day -1. Subjects should be instructed not to drink alcohol within 12 hours of the screening assessment.
* Intake of alcohol within 72 hours prior to study drug administration or intake of grapefruit or Seville oranges within 7 days prior to the administration of study drug.
* Strenuous physical exercise within 48 hours prior to study drug administration.
* Administration of any over-the-counter medication, dietary supplements, or vitamins within 7 days prior to study drug administration. Excluded from this list is nondaily use of acetaminophen at doses of ≤2 grams over a 24-hour period.
* Administration of prescription drugs or herbal supplements within 14 days prior to study drug administration.

  -.Exposure to any investigational agent within 30 days prior to the Screening Visit.
* Any current medical illness, signs, or symptoms that, in the investigator's opinion, could adversely affect subject safety or study integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be the number and severity of treatment emergent adverse events (TEAEs) following single doses of EC-18 and placebo. | 30 days

SECONDARY OUTCOMES:
To determine the composite pharmacokinetic (PK) parameters of EC-18 following sngle oral doses. AUC0-t, AUC0-24, Cmax, Tmax, 48-hour time period. | Predose [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 hours post dose
  AUC0-t: Area under the plasma drug concentration versus time curve from time zero to time t; AUC0-24: Area under the plasma concentration versus time curve from time zero to 24 hours after dosing, Cmax: Maximum observed plasma drug concentration; Tmax: Time of maximum drug concentration

OTHER OUTCOMES:
To determine the pharmacodynamic effects of EC-18 on circulating leukocyte cell counts. | Day 5 after dosing.
To determine the pharmacodynamic effects of EC-18 on red blood cell counts. | Day 5 after dosing.
To determine the pharmacodynamic effects of EC-18 on reticulocyte counts. | Day 5 after dosing.
To determine the pharmacodynamic effects of EC-18 on platelet counts. | Day 5 after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Treva W Tyson, MD, Principal Investigator — Wake Research Associates
Locations (1):
- Carolina Phase I Clinical Research, Raleigh, North Carolina, United States